CLINICAL TRIAL: NCT03589183
Title: Discovery of Gut Microbial Signatures in Inflammatory Bowel Disease
Brief Title: Gut Microbiome in Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Professor, Kyunghee University Medical Center
Other Study IDs: IBD library_2018
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Gut Microbiome; Ulcerative colitis; Crohn disease; Multi-omics; Psychometrics; anxiety; depression
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (whole blood and serum), fecal and mucosal sample from each study subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory condition for gastrointestinal tract. There have been numerous studies to reveal dysbiosis of fecal/mucosal microbiome composition in IBD patients but actual trend of dysbiosis is strikingly different among patient's ethnicity.

In this background, the investigators have composed a prospective cohort of Korean IBD patients in a large academic referral IBD center. Using an integrated multi-omics bioinformatic analysis, the investigators aim to explore gut microbial signatures along with distinct clinical/genetic features, and their potential interplay in patients with IBD.

DETAILED DESCRIPTION:
This prospective cohort study aims to build a gut microbiome library for Korean IBD patients, and also aims to explore gut microbial signatures along with distinct clinical/genetic features and their potential interplay using the investigator's multi-omics analysis platform.

After signing the informed consent, various biological samples (fecal, mucosal and blood samples) as well as comprehensive clinical data (including psychometric evaluations using patient survey) will be obtained from patients periodically.

The multi-omics investigations will comprise: metagenomics (16s RNA sequencing and whole metagenomic sequecing), metabolomics, human genomics (genome-wide SNP data, whole exome and genome sequencing), transcriptomics, proteomics, epigenetics and single-cell multi-omics analysis. In vitro and in vivo study using fecal samples will be conducted.

In brief, after extracting the DNA from blood samples, whole genome sequencing will be performed and data will be compared with the previously reported variances. Novel variances or incidence of specific variances will be measured. Fecal sample will be collected and microbiome composition of each study subjects will be analyzed. Fecal microbial diversity will be measured from sequencing data of 16S ribosomal RNA which is highly preserved area of genetic information amongst microorganisms. Colonic mucosal sample will be collected when routine endoscopic surveillance is planned. Sample will be collected from diseased and normal mucosal altogether for analysis. Microbial diversity will be measured from 16S RNA sequencing data of the samples.

The multi-omics data will be analyzed with comprehensive clinical metadata using an integrated bioinformatics analysis platform. Clinical data include demographics, disease characteristics and variouis patient-reported outomes data (including health-related quality of life, anxiety, depression and others). Patient-reported outcomes data will be collected using validated questionnaires periodically.

Data from basic analysis will be re-explore in terms of inter-individual difference, difference between disease characteristics (such as disease phenotype, type of medical treatment and serologic markers), difference between psychosocial characteristics (such as the presence of anxiety or depression and quality of life) and etc. In addition, data from basic analysis will be used as the reference for the Korean IBD patient and it will be compared with other data obtained from the "different ethnicity" or "healthy" Korean population.

In conclusion, this long term, large-scale prospective study will provide a platform for studying a field of translational medicine to reveal hidden signatures of gut microbiome underlying IBD and to identify potential biological markers in IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of inflammatory bowel disease, including ulcerative colitis and Crohn disease

Exclusion Criteria:

* Person with history of using antibiotics or probiotics within previous 2 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are planned to study all patients with established diagnosis of IBD (Crohn disease or ulcerative colitis) registered in single tertiary referral IBD center (KyungHee University Medical Center).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Composition and diversity of gut microbiome | Up to 10 years
  Fecal and/or intestinal mucosal samples are obtained from enrolled subjects for metagenomic sequencing. After extracting fecal or mucosal DNA, microbial composition and diversity are measured from 16sRNA high-throuput sequencing or Shotgun method. Data are compared across different disease phenotypes, such as types of disease (ulcrerative colitis versus Crohn's disease), type of treatment and the presence of psychological disorders (anxiety/depression).

SECONDARY OUTCOMES:
Taxonomic profiling of gut microbiome | Up to 10 years
  Fecal and/or intestinal mucosal samples are obtained from enrolled subjects for metagenomic sequencing. After extracting fecal or mucosal DNA, taxonomic profiles associated with inflammatory bowel diseases and different disease phenotypes are analyzed from 16sRNA high-throuput sequencing or Shotgun method.
Finding of single nucleotide polymorphisms (SNPs) | Up to 10 years
  Blood samples are obatined from enrolled subjects for genome-wide microarray. After extracting DNA, SNPs related to inflammatory bowel diseases and different disease phenotypes are explored (Genome-wide association study [GWAS] statistical significance threshold, P < 5.00*E-08).
Finding of serologic biomarkers | Up to 10 years
  Blood samples are obatined from enrolled subjects for proteomic analysis. Serologic biomakers implicating in inflammatory bowel diseases and disease phenotypes are explored.
Correlation between host genotyping and gut microbiome | Up to 10 years
  Blood samples are obatined from enrolled subjects for genome-wide microarray. After extracting DNA, SNPs related to inflammatory bowel diseases and different disease phenotypes are explored (Genome-wide association study [GWAS] statistical significance threshold, P < 5.00*E-08). Fecal and/or intestinal mucosal samples are obtained from enrolled subjects for metagenomic sequencing. After extracting fecal or mucosal DNA, taxonomic profiles associated with inflammatory bowel diseases and different disease phenotypes are analyzed from 16sRNA high-throuput sequencing or Shotgun method. Taxonomic composition of gut microbiome are compared according to the sequecing data of host genomes .
Liquid biopsy biosignatures assessed by single cell RNA-Seq | Up to 10 years
  Blood and intestinal mucosal biopsy samples are obtained from enrolled subjects, particularly those treated with biological drugs or small molecues for single cell analysis (RNA-Seq). Data obtained from single cell analysis will be compared across different time frame (for example, before versus after specific treatment) and across differnt disease phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Jong Kim, MD PhD, Principal Investigator — KyungHee University Hospital; Chang Kyun Lee, MD PhD, Principal Investigator — KyungHee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
After publishing the results, any data sharing request from other researchers will be positively considered. But extent of sharing is not decided yet.

REFERENCES:
- [Background] Wellcome Trust Case Control Consortium. Genome-wide association study of 14,000 cases of seven common diseases and 3,000 shared controls. Nature. 2007 Jun 7;447(7145):661-78. doi: 10.1038/nature05911. PMID 17554300
- [Background] Thia KT, Loftus EV Jr, Sandborn WJ, Yang SK. An update on the epidemiology of inflammatory bowel disease in Asia. Am J Gastroenterol. 2008 Dec;103(12):3167-82. doi: 10.1111/j.1572-0241.2008.02158.x. PMID 19086963
- [Background] Nishida A, Inoue R, Inatomi O, Bamba S, Naito Y, Andoh A. Gut microbiota in the pathogenesis of inflammatory bowel disease. Clin J Gastroenterol. 2018 Feb;11(1):1-10. doi: 10.1007/s12328-017-0813-5. Epub 2017 Dec 29. PMID 29285689
- [Background] Huang H, Vangay P, McKinlay CE, Knights D. Multi-omics analysis of inflammatory bowel disease. Immunol Lett. 2014 Dec;162(2 Pt A):62-8. doi: 10.1016/j.imlet.2014.07.014. Epub 2014 Aug 15. PMID 25131220